CLINICAL TRIAL: NCT07404020
Title: AI-Powered OSCE Coaching in Improving Infertility Counseling Skills: A Randomized Controlled Study in Nursing Students
Brief Title: AI-Powered OSCE Coaching in Improving Infertility Counseling Skills in Nursing Students
Acronym: AI-OSCE-Infert
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, GÜLESER ADA, Assistant Professor, Bartın Unıversity
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BARU-SBF-OSCE-AI-2026
Record Dates: First submitted 2026-02-01; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Infertility Counseling; Communication Skills
Keywords: Infertility counseling; nursing education; artificial intelligence; OSCE; therapeutic communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Participants receive generative AI-supported OSCE coaching using structured infertility counseling scenarios with automated feedback and deliberate practice.
  Interventions: Behavioral: AI-Powered OSCE Coaching
- control (No Intervention): No intervention will be made to the control group. Only measurements will be made on parallel dates with the experimental group.

INTERVENTIONS:
Behavioral: AI-Powered OSCE Coaching — Participants receive a generative artificial intelligence-supported OSCE coaching intervention designed to improve infertility counseling communication and empathy skills. The intervention consists of 6-8 structured micro-scenarios reflecting common infertility counseling situations. For each scenario, participants provide written counseling responses, which are analyzed by the AI system based on therapeutic communication and empathy principles. Automated, structured feedback is provided, allowing participants to revise and repeat responses in a deliberate practice cycle. The intervention is delivered individually and does not involve real patients.
  Arms: Experimental group

SUMMARY:
This randomized controlled experimental study aims to evaluate the effectiveness of a generative artificial intelligence-based "OSCE Coach" in improving infertility counseling communication and empathy skills among nursing students. The study will be conducted with undergraduate nursing students at Bartın University Faculty of Health Sciences and follows a two-group pretest-posttest design.

A total of 96 students will be randomly assigned to either the intervention group or the control group using computer-generated randomization. The intervention group will participate in an AI-powered OSCE coaching simulation consisting of 6-8 infertility counseling micro-scenarios, incorporating structured feedback and deliberate practice cycles. The control group will receive conventional infertility counseling education using standard teaching methods.

Outcomes will be assessed using the Therapeutic Communication Skills Scale for Nursing Students, the Jefferson Scale of Empathy for Nursing Students, and a rubric-based infertility counseling communication performance assessment based on the Kalamazoo Consensus Statement. Performance evaluations will be conducted via standardized virtual patient interviews and scored by two blinded independent raters.

Data will be analyzed using ANCOVA to assess intervention effects while controlling for baseline scores. This study aims to contribute evidence on the effectiveness of AI-supported OSCE coaching in enhancing communication and empathy skills in nursing education.

DETAILED DESCRIPTION:
This study is designed as a two-group, randomized controlled experimental trial with a pretest-posttest design to evaluate the effectiveness of a generative artificial intelligence-based "OSCE Coach" in improving infertility counseling communication and empathy skills among nursing students. The study will be conducted at Bartın University Faculty of Health Sciences, Department of Nursing, following approval from the Bartın University Social and Humanities Ethics Committee and in accordance with the principles of the Declaration of Helsinki.

The study population will consist of undergraduate nursing students who are actively enrolled in the infertility nursing course and have successfully completed the women's health and diseases nursing course. Eligible participants who provide written informed consent will be randomly assigned to either the intervention group or the control group using a computer-generated randomization sequence. Allocation will be performed by an independent individual not involved in data collection or analysis. Due to the nature of the educational intervention, participant blinding will not be possible; however, outcome assessors evaluating OSCE performance will be blinded to group allocation.

The intervention group will receive training through a generative artificial intelligence-based "OSCE Coach" designed to support deliberate practice in infertility counseling communication. The intervention consists of 6-8 structured micro-scenarios reflecting common and challenging infertility counseling situations, including establishing rapport, psychosocial assessment, managing emotional reactions, addressing partner-related concerns, responding to social stigma, providing clear information, delivering difficult news, and closing the counseling session. In each scenario, participants will provide written counseling responses, which will be analyzed by the AI system based on therapeutic communication and empathy principles. Structured, rubric-based feedback will be provided, allowing participants to revise and repeat their responses in a deliberate practice cycle.

The control group will receive conventional infertility counseling education delivered through standard teaching methods, including lectures, written case discussions, and review of example counseling dialogues. The duration and overall educational workload of the control condition will be matched to that of the intervention group to ensure comparability between groups. No AI-supported simulation or interactive feedback will be used in the control group.

Outcome assessment will be conducted using validated self-report scales and a standardized performance-based evaluation. Therapeutic communication skills will be measured using the Therapeutic Communication Skills Scale for Nursing Students, and empathy levels will be assessed using the Jefferson Scale of Empathy for Nursing Students. Counseling performance will be evaluated through standardized virtual patient interviews conducted in an examination-mode simulation environment. All participants will complete the same virtual patient scenario under identical conditions. Performances will be scored independently by two trained evaluators using a rubric developed based on the Kalamazoo Consensus Statement. Evaluators will be blinded to participants' group assignments, and inter-rater reliability will be assessed using the intraclass correlation coefficient.

Pretest assessments will be conducted prior to the educational intervention, and posttest assessments will be completed after the intervention period. Data will be analyzed using appropriate parametric or non-parametric statistical methods based on data distribution. Analysis of covariance (ANCOVA) will be used to evaluate intervention effects while controlling for baseline scores. Effect sizes will be calculated, and statistical significance will be set at p < 0.05.

All participant data will be anonymized using unique identification codes. Only the research team will have access to the data, which will be stored securely and used solely for scientific purposes. Participants will have the right to withdraw from the study at any time without penalty. Upon completion of the study, students in the control group will be offered optional access to the AI-based OSCE coaching system in line with ethical considerations.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate nursing students enrolled at Bartın University Faculty of Health Sciences
* Successfully completed the Women's Health and Diseases Nursing course (minimum passing grade)
* Currently enrolled in the infertility nursing course
* Able to read and understand Turkish
* Willing to participate and provide written informed consent

Exclusion Criteria:

* Students who do not complete the educational intervention
* Students who do not complete pretest or posttest assessments
* Students with prior formal training in AI-supported OSCE or similar simulation-based coaching programs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Infertility Counseling Communication Performance | Post-intervention (immediately after completion of the AI-powered OSCE coaching or conventional training)
  Counseling communication performance assessed through standardized virtual patient interviews using a rubric-based evaluation tool developed based on the Kalamazoo Consensus Statement. Performances are independently scored by two blinded evaluators, and the average score is used for analysis.

SECONDARY OUTCOMES:
Therapeutic Communication Skills | Baseline (prior to intervention) and post-intervention (immediately after completion of the intervention)
  Measured using the Therapeutic Communication Skills Scale for Nursing Students. Total scores range from 16 to 112, with higher scores indicating better therapeutic communication skills.
Clinical Empathy Level | Baseline (prior to intervention) and post-intervention (immediately after completion of the intervention)
  Measured using the Jefferson Scale of Empathy for Nursing Students. Total scores range from 18 to 126, with higher scores indicating higher empathy levels.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru CİRBAN EKREM, PhD, Study Director — Bartın Unıversity; Harun İlçioğlu, PhD, Principal Investigator — Kastamonu University; Kevser İlçioğlu, PhD, Principal Investigator — sakarya üniversity
Locations (1):
- Bartın University, Merkez, Bartın, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No